CLINICAL TRIAL: NCT04373759
Title: Cardiac Arrest Incidence and Outcome Among Patient With COVID-19 Pneumonia in French ICUs
Brief Title: Cardiac Arrest Incidence and Outcome Among Patients With COVID-19 in French ICUs
Acronym: ACICOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-CHITS-004
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Sars-CoV2; Covid-19
Keywords: novel coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Out-of-hospital cardiac arrest; In-hospital cardiac arrest; unexpected cardiac arrest; Intensive care unit
MeSH Terms: conditions — COVID-19; Out-of-Hospital Cardiac Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unexpected in-intensive care unit cardiac arrest patients: ICUCA Patients admitted in intensive care unit for a confirmed COVID-19 and presenting an unexpected in-intensive care unit cardiac arrest
  Interventions: Other: Cardiopulmonary resuscitation; Other: Modified Rankin score
- In-hospital cardiac arrest patients: IHCA Patients admitted in intensive care unit for an in-hospital cardiac arrest with a confirmed Covid-19
  Interventions: Other: Modified Rankin score
- Out-of-hospital cardiac arrest: OHCA Patients admitted in intensive care unit for an out-hospital cardiac arrest with a confirmed Covid-19
  Interventions: Other: Modified Rankin score

INTERVENTIONS:
Other: Cardiopulmonary resuscitation — Cardiopulmonary resuscitation
  Groups: Unexpected in-intensive care unit cardiac arrest patients
Other: Modified Rankin score — 0 - no symptoms at all
  1. - no significant disability despite symptoms; able to carry out all usual duties and activities
  2. - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. - Moderate disability; requiring some help, but able to walk without assistance
  4. - Moderately severe disability; unable to walk and attend to bodily needs without assistance
  5. - Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. - Dead

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is responsible for the novel coronavirus disease 2019 (COVID-19) pandemic. Among COVID-19 complications, in-hospital cardiac arrest (IHCA) was reported with a very poor outcome in a retrospective single-center study (0,7% of 30 days survival with good neurological outcome among IHCA patients with a resuscitation attempt), related to its natural course and management. The incidence of unexpected in-ICU cardiac arrest (ICUCA) due to COVID-19 is still unknown. Additionally, outcome of COVID-19 patients admitted in ICU for an out-of-hospital cardiac arrest (OHCA) is also undescribed.

The objective this study is :

* to report the incidence of ICUCA among patients hospitalized in French ICU for COVID-19.
* to report morbidity and mortality among COVID-19 patients admitted alive in ICU for an OHCA or an IHCA.

The secondary objective is to assess outcome and identify risk factors of ICUCA occurrence among patients admitted for COVID-19.

DETAILED DESCRIPTION:
Retrospective and prospective multicentric observational registry in French intensive care units (ICU) including all consecutive adult patients admitted in ICU with a documented SARS-CoV-2 disease :

* For an out-of-hospital or an in-hospital cardiac arrest (OHCA and IHCA respectively)
* Or presenting an unexpected in-ICU cardiac arrest (ICUCA) Patients characteristics, cardiac arrest history and patients outcome will be recorded according to Utstein recommendations.

Patients presenting an expected cardiac arrest in ICU related to withdrawal of life sustaining therapies (WLST) will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in intensive care unit with a documented SARS-CoV-2 disease
* For an out-of-hospital or an in-hospital cardiac arrest
* Or an in-hospital cardiac arrest
* Or presenting an unexpected in-intensive care unit cardiac arrest

Exclusion Criteria:

* Age under 18 y.o
* Expected in-intensive care unit cardiac arrest related to withdrawal of life sustaining therapies.
* Withdrawal of patient or next-of-kin informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients admitted in intensive care unit with a documented SARS-CoV-2 disease
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of unexpected cardiac arrest | 7 months
  Percentage of unexpected in-intensive care unit cardiac arrest among COVID-19 patients admitted to intensive care unit

SECONDARY OUTCOMES:
Charlson score | 7 months
  Diabetes, hypertension, smoking, dyslipidemia, coronary artery disease, chronic respiratory insufficiency, chronic heart failure, chronic renal insufficiency, chronic hepatic insufficiency, chronic neurological disease, cancer, malignant hemopathy. Charlson score's minimum and maximum values are 0 and 40 respectively, the lowest score corresponds to a better outcome.
Organ failure score at ICU admission and/or before unexpected in-ICU cardiac arrest | 7 months
  Respiratory failure, neurological impairment, circulatory failure, hepatic failure, haematological failure, renal failure. Sofa score's minimum and maximum values are 0 and 24, the lowest score corresponds to a better outcome
Etiology retained to explain cardiac arrest occurrence | 7 months
  Cardiac origin; Respiratory origin; Metabolic origin; unknown origin
Modified Rankin score (mRS) at ICU discharge, at hospital discharge and at 3 months | 3 months
  0 - no symptoms at all
  1. - no significant disability despite symptoms; able to carry out all usual duties and activities
  2. - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. - Moderate disability; requiring some help, but able to walk without assistance
  4. - Moderately severe disability; unable to walk and attend to bodily needs without assistance
  5. - Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. - Dead

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Chelly, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (36):
- France (35):
  - CHU Caen, Caen, Calvados
  - Hôpital Privé St Martin, Caen, Calvados
  - CH Angoulème, Angoulême, Charente
  - CH Brive, Brive-la-Gaillarde, Corrèze
  - CHU Dijon, Dijon, Côte-d'Or
  - CH Etampes, Étampes, Essonne
  - CHU Antoine Béclère AP-HP, Clamart, Haut-de-Seine
  - CHU Ambroise Paré AP-HP, Boulogne-Billancourt, Hauts-de-Seine
  - CH Louis Mourier AP-HP, Colombes, Hauts-de-Seine
  - CHU Montpellier, Montpellier, Hérault
  - CHU Felix Guyon, Saint-Denis, La Reunion
  - CHR Orléans, Orléans, Loiret
  - CH Cahors, Cahors, Lot
  - CHRU Roger Salengro, Lille, Nord
  - CH Bethune, Beuvry, Pas-de-Calais
  - CH Lens, Lens, Pas-de-Calais
  - Grand Hôpital de l'Est Francilien, Jossigny, Seine-et-Marne
  - CHU Meaux, Meaux, Seine-et-Marne
  - Groupe Hospitalier Sud Ile de France, Melun, Seine-et-Marne
  - CHU Rouen, Rouen, Seine-Maritime
  - CHU Amiens Picardie, Amiens, Somme
  - Hôpital Nord Franche Comté, Trévenans, Territoire De Belfort
  - CH Argenteuil, Argenteuil, Val-d'Oise
  - CHU Henri Mondor AP-HP, Créteil, Val-de-Marne
  - CHU Kremlin Bicêtre, Le Kremlin-Bicêtre, Val-de-Marne
  - CH de la Dracénie, Draguignan, Var
  - CHI Frejus St Raphael, Fréjus, Var
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var
  - CH Versailles, Le Chesnay, Yvelines
  - CHU Lariboisière AP-HP, Paris, Île-de-France Region
  - CHU Saint Louis AP-HP, Paris, Île-de-France Region
  - CHU St Antoine, Paris, Île-de-France Region
  - Groupe Hospitalier Saint Joseph, Paris, Île-de-France Region
  - CHU Necker Enfants Malades, Paris, Île-de-France Region
  - CHU Pitié Salpétrière, Paris, Île-de-France Region
- CHU Martinique - Fort de France, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Leloup M, Briatte I, Langlois A, Cariou A, Lesieur O; ACIR study group. Unexpected cardiac arrests occurring inside the ICU: outcomes of a French prospective multicenter study. Intensive Care Med. 2020 May;46(5):1005-1015. doi: 10.1007/s00134-020-05992-w. Epub 2020 Mar 9. PMID 32152653
- [Background] Bansal M. Cardiovascular disease and COVID-19. Diabetes Metab Syndr. 2020 May-Jun;14(3):247-250. doi: 10.1016/j.dsx.2020.03.013. Epub 2020 Mar 25. PMID 32247212
- [Background] Chen C, Zhou Y, Wang DW. SARS-CoV-2: a potential novel etiology of fulminant myocarditis. Herz. 2020 May;45(3):230-232. doi: 10.1007/s00059-020-04909-z. No abstract available. PMID 32140732
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Madjid M, Safavi-Naeini P, Solomon SD, Vardeny O. Potential Effects of Coronaviruses on the Cardiovascular System: A Review. JAMA Cardiol. 2020 Jul 1;5(7):831-840. doi: 10.1001/jamacardio.2020.1286. PMID 32219363
- [Background] Wu CI, Postema PG, Arbelo E, Behr ER, Bezzina CR, Napolitano C, Robyns T, Probst V, Schulze-Bahr E, Remme CA, Wilde AAM. SARS-CoV-2, COVID-19, and inherited arrhythmia syndromes. Heart Rhythm. 2020 Sep;17(9):1456-1462. doi: 10.1016/j.hrthm.2020.03.024. Epub 2020 Mar 31. PMID 32244059
- [Background] Shao F, Xu S, Ma X, Xu Z, Lyu J, Ng M, Cui H, Yu C, Zhang Q, Sun P, Tang Z. In-hospital cardiac arrest outcomes among patients with COVID-19 pneumonia in Wuhan, China. Resuscitation. 2020 Jun;151:18-23. doi: 10.1016/j.resuscitation.2020.04.005. Epub 2020 Apr 10. PMID 32283117
- [Background] Chan PS, Berg RA, Nadkarni VM. Code Blue During the COVID-19 Pandemic. Circ Cardiovasc Qual Outcomes. 2020 May;13(5):e006779. doi: 10.1161/CIRCOUTCOMES.120.006779. Epub 2020 Apr 7. PMID 32255661
- [Background] Mahase E, Kmietowicz Z. Covid-19: Doctors are told not to perform CPR on patients in cardiac arrest. BMJ. 2020 Mar 29;368:m1282. doi: 10.1136/bmj.m1282. No abstract available. PMID 32224494
- [Background] Perkins GD, Jacobs IG, Nadkarni VM, Berg RA, Bhanji F, Biarent D, Bossaert LL, Brett SJ, Chamberlain D, de Caen AR, Deakin CD, Finn JC, Grasner JT, Hazinski MF, Iwami T, Koster RW, Lim SH, Ma MH, McNally BF, Morley PT, Morrison LJ, Monsieurs KG, Montgomery W, Nichol G, Okada K, Ong ME, Travers AH, Nolan JP; Utstein Collaborators. Cardiac Arrest and Cardiopulmonary Resuscitation Outcome Reports: Update of the Utstein Resuscitation Registry Templates for Out-of-Hospital Cardiac Arrest: A Statement for Healthcare Professionals From a Task Force of the International Liaison Committee on Resuscitation (American Heart Association, European Resuscitation Council, Australian and New Zealand Council on Resuscitation, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa, Resuscitation Council of Asia); and the American Heart Association Emergency Cardiovascular Care Committee and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. Resuscitation. 2015 Nov;96:328-40. doi: 10.1016/j.resuscitation.2014.11.002. Epub 2014 Nov 11. PMID 25438254
- [Result] Chelly J, Plantefeve G, Kamel T, Bruel C, Nseir S, Lai C, Cirillo G, Skripkina E, Ehrminger S, Berdaguer-Ferrari FD, Le Marec J, Paul M, Autret A, Deye N; ACICOVID-19 study group. Incidence, clinical characteristics, and outcome after unexpected cardiac arrest among critically ill adults with COVID-19: insight from the multicenter prospective ACICOVID-19 registry. Ann Intensive Care. 2021 Nov 13;11(1):155. doi: 10.1186/s13613-021-00945-y. PMID 34773516